CLINICAL TRIAL: NCT03089632
Title: The Effect of Gluten-free Diet on Upper Gastrointestinal Symptoms in Type 1 Diabetic Patients With Dyspepsia-like Symptoms
Brief Title: The Effect of Gluten-free Diet in Type 1 Diabetics With Dyspepsia Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM1 and GFD_01
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 1; Gastroparesis; Dyspepsia; Gluten Sensitivity
Keywords: gluten-free diet; gluten sensitivity; dyspepsia; diabetes mellitus, type 1; gastroparesis; motility
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Gastroparesis; Dyspepsia; Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Before and after clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluten-free diet (Experimental): All patients will follow a strict gluten-free diet for 1 month. Measurement will be conducted at baseline and after the intervention.
  Interventions: Other: Gluten-free diet

INTERVENTIONS:
Other: Gluten-free diet — One-month gluten-free diet

SUMMARY:
Patients with type-1 diabetes are more susceptible to motility-related upper gastrointestinal symptoms. Dietary interventions are one of the treatment pillars for these symptoms. Many gastrointestinal conditions other than celiac disease, are being increasingly treated with gluten-free diet (GFD). The role of GFD in non-celiac type-1 diabetic patients with dyspepsia-like symptoms has not been assessed before. In this study, type 1 diabetes patients with concomitant upper gastrointestinal symptoms will be asked to follow a 1-month GFD to assess changes in upper gastrointestinal symptoms and gastroduodenal motility before and after the dietary intervention.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a complex and heterogeneous disease that is associated with poor outcomes. In studies from referral centers, 50-65% of diabetics reported dyspeptic symptoms. In addition, approximately 50% of type 1 DM (T1DM) patients, especially those with longstanding disease, have evidence of delayed gastric emptying.

Dietary modification is one of the treatment pillars for patients with dyspeptic symptoms. Further, many individuals in which both symptoms and motility abnormalities improve after a GFD have positive anti-gliadin antibodies (AGA), which reinforces the role of gluten-induced inflammation/immune activation as a possible cause of motility abnormalities and related symptoms.

Ameliorating UGI symptoms is not only pivotal for improving the quality of life of diabetic GP patients, but the improvement in gastroduodenal motility is also needed for a more predictable glycemic response. In non-celiac T1DM patients, the role of the GFD in symptom improvement, gastroduodenal motility and glycemic control has never been assessed.

The overall aim of the present study is to improve the knowledge about the role of dietary interventions as non-pharmacological treatments for upper-gastrointestinal symptoms and underlying motility abnormalities in patients with type 1 diabetes. This will be a non-randomized, open label, before and after trial of a 1-month GFD in non-celiac type 1 diabetics to assess symptomatic, motility and glycemic response changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (18-75 years) with type 1 diabetes diagnosis and no history of celiac disease, that complain of upper gastrointestinal symptoms (early satiety, postprandial fullness, bloating, abdominal swelling, nausea, vomiting, and retching) will be invited to participate.

Exclusion Criteria:

* Patients with very severe symptoms of gastroparesis that require specialized nutritional therapy or surgical treatment;
* Pregnant women;
* Patients with concomitant diseases/treatments that can alter gastrointestinal motility and concomitant severe systemic diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in upper gastrointestinal symptoms assessed by the Leeds short-form questionnaire (SF-LDQ) | 1 month
  Difference in upper gastrointestinal symptoms' severity (before and after the dietary intervention) assessed by the Leeds short-form questionnaire (SF-LDQ)
Changes in upper gastrointestinal symptoms assessed by the Gastroparesis Cardinal Symptoms Index (GCSI) | 1 month
  Difference in upper gastrointestinal symptoms' severity (before and after the dietary intervention) assessed by the Gastroparesis Cardinal Symptoms Index (GCSI).

SECONDARY OUTCOMES:
Changes in gastric emptying determined by gastric scintigraphy. | 1 month
  Difference in gastric emptying (before and after the intervention) determined by gastric scintigraphy.
Changes in gastro-duodenal motility assessed by videofluoroscopy | 1 month
  Differences in gastro-duodenal contraction patterns (before and after the intervention) assessed by videofluoroscopy.
Changes in glycemic control assessed by continuous glucose monitoring | 1 month
  Differences in continous glucose monitoring (before and after the intervention) assessed by 6-day continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Bercik, MD, PhD, Principal Investigator — McMaster University, Department of Medicine, Division of Gastroenterology
Locations (1):
- McMaster Health Sciences Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No